CLINICAL TRIAL: NCT05590624
Title: Elucidating the Metabolic Impact of Isocaloric, Controlled, Mediterranean-Type Diets in Treatment-Naïve Men With Prostate Cancer on Active Surveillance (DINE Study)
Brief Title: Metabolic Impact of Prospective Controlled Mediterranean Type Diets on Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CASE4822
Record Dates: First submitted 2022-09-23; First posted 2022-10-21 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Mediterranean-type Diets
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two arms which only differ in the order they will receive the two dietary interventions [Lower Carbohydrate (LC) and Low Fat (LF)]. All dietary interventions are on a Mediterranean foundation and are opposite in carbohydrate and fat content.
  Arm 1 [n=15 with confirmed PCa diagnosis and candidate for Active Surveillance (AS) per Standard of Care (SOC)]: Dietary Intervention #1=Low Fat (LF) Mediterranean. Dietary Intervention #2=Lower Carbohydrate (LC) Mediterranean
  Arm 2 (n=15 with confirmed PCa diagnosis and candidate for AS per SOC): Dietary Intervention #1=LC Mediterranean. Dietary Intervention #2=LF Mediterranean
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean-type Diet(s)-Arm 1 (Experimental): Diet randomization occurs two weeks prior to the Standard of Care (SOC) diagnostic biopsy. If patient is randomized to Arm 1, they will receive Low Fat (LF) Mediterranean Diet first. The results of the diagnostic biopsy determines how the patient will proceed on the trial. If there is a confirmed Prostate Cancer (PCa) diagnosis AND is a candidate for Active Surveillance (AS) per SOC, then patient will undergo a washout period and cross-over to the Lower Carbohydrate (LC) Mediterranean Diet two weeks prior to the SOC confirmatory biopsy. A long-term follow-up (LTFU) visit will occur 3 months after the second dietary intervention has concluded. If patient does not have PCa or is not placed on AS, then they will only have the first dietary intervention and a LTFU visit 3 months after
  Interventions: Other: Lower-Carbohydrate Med-t-Diet; Other: Low-Fat Med-t-Diet
- Mediterranean-type Diet(s)-Arm 2 (Experimental): Diet randomization occurs two weeks prior to the Standard of Care (SOC) diagnostic biopsy. If patient is randomized to Arm 2, they will receive Lower Carbohydrate (LC) Mediterranean Diet first. The results of the diagnostic biopsy determines how the patient will proceed on the trial. If there is a confirmed Prostate Cancer (PCa) diagnosis AND is a candidate for Active Surveillance (AS) per SOC, then patient will undergo a washout period and cross-over to the Low Fat (LF) Mediterranean Diet two weeks prior to the SOC confirmatory biopsy. A long-term follow-up (LTFU) visit will occur 3 months after the second dietary intervention has concluded. If patient does not have PCa or is not placed on AS, then they will only have the first dietary intervention and a LTFU visit 3 months after.
  Interventions: Other: Lower-Carbohydrate Med-t-Diet; Other: Low-Fat Med-t-Diet

INTERVENTIONS:
Other: Lower-Carbohydrate Med-t-Diet — Diet will focus on including:
  * Lean protein sources
  * High-quality fat
  * High-quality carbohydrate sources that are rich in fiber
  * Nuts and seeds
  Diet will focus on limiting:
  * Refined sugars
  * High glycemic carbohydrates
  * Seed oils that may cause inflammation
  Diet Composition: 45% fats, 35% carbs, 20% protein
Other: Low-Fat Med-t-Diet — Diet will focus on including:
  * Lean protein sources
  * High-quality fat
  * High-quality carbohydrate sources that are rich in fiber
  * Nuts and seeds
  Diet will focus on limiting:
  * Refined sugars
  * High glycemic carbohydrates
  * Seed oils that may cause inflammation
  Diet Composition: 70% carbs, 20% protein, 10% fat

SUMMARY:
The purpose of this study is to examine the impact of Mediterranean-type diets on the metabolism of men with localized prostate cancer.

The optimal diet for men with a suspected diagnosis of Prostate Cancer (PCa) is currently unknown. More specifically, the suggested benefits of low carbohydrate and low fat diets in PCa are not determined.

DETAILED DESCRIPTION:
Primary Objective

-Evaluate the impact of Mediterranean diets (Med-t-Diets) on non-malignant prostate tissue metabolism

Secondary Objectives

* Evaluate the impact of Med-t-Diets on host metabolism
* Evaluate the impact of Med-t-Diets on systemic biomarkers after consuming Med-t-Diets
* Evaluate the impact of Med-t-Diets on the microbiome and dietary behavior and compliance after consuming Med-t-Diets

ELIGIBILITY:
Inclusion Criteria:

* Males ≥18 years old
* High suspicion of prostate cancer (PCa) per urologist's clinical evaluation
* BMI >18.5
* No prior PCa diagnosis or hormonal therapy (-ies)
* Ability to read, write, speak, and understand English
* Ability to provide informed consent
* Candidate for and elects active surveillance (AS) if diagnostic biopsy is positive
* Willingness to consume provided dietary interventions
* Adequate organ and marrow function: White blood cell count (WBC) ≥2,500/mcL, Absolute neutrophil count (ANC) ≥1,500/mcL, Platelets ≥100,000/mcL, Hemoglobin ≥9 g/dL (transfusions permitted), Total bilirubin ≤1.5 x the institutional upper limit of normal (ULN) (for subjects with Gilbert's disease ≤3.0 mg/dL), Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) ≤2.5 x institutional ULN, Creatinine clearance ≥51 ml/min as defined by Cockcroft-Gault equation

Exclusion Criteria:

* Currently consuming a Mediterranean, lower carbohydrate, ketogenic, vegan, vegetarian, high fiber diet (14g fiber > per 1,000 Calories) and/or any supplements (including herbal), vitamins, minerals, that would interfere with diets being tested in the study as determined by dietitian and/or investigators.
* Previous intolerability to fiber-rich diets
* Colitis, Irritable Bowel Syndrome, or other gastrointestinal condition per clinician discretion
* Unwilling to undergo transperineal PCa biopsies
* Food allergies or other major dietary restrictions
* Receiving active medical treatment for Type I or Type II diabetes mellitus
* Prior antibiotic usage (i.e. within last 30 days) at time of consent
* Recent weight loss (both intentional and unintentional) as defined by 5%+ body weight in the last 30 days
* Undergone any type of weight loss surgery
* Any medical contraindications as determined by investigators
* High risk as defined by PSA≥20 and/or PI-RADS 5 lesion as per clinician evaluation
* History of diabetic ketoacidosis
* Gout
* Patients that are immunosuppressed (transplant history, on immunosuppression, etc.) as per clinician discretion
* Recent (within last 30 days) device implant/joint requiring antibiotics as per clinician determination
* Prior history of prostate biopsy infection
* Uncontrolled hypertension as defined by blood pressure greater than 140/80 (with or without medication)
* Gallbladder removed or plan to remove per clinician evaluation
* Other malignancies actively receiving systemic treatment as per clinician evaluation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of Med-t-Diets on non-malignant prostate tissue metabolism | Change from diagnostic biopsy (Week 2) at confirmatory biopsy
  Change in non-malignant prostate tissue metabolomics using mass spectrometry to assess differences in ions/metabolites and corresponding metabolic pathways after different dietary interventions expressed as a fold-change. As an exploratory study, metabolomics will be untargeted and as such is not run with a standard curve and does not have a unit of measure.

SECONDARY OUTCOMES:
Changes in blood metabolomics | Change from baseline at two weeks on diet
  Change in blood metabolomics using mass spectrometry to assess differences in ions/metabolites and corresponding metabolic pathways after different dietary interventions expressed as a fold-change. As an exploratory study, metabolomics will be untargeted and as such is not run with a standard curve and does not have a unit of measure
Changes in energy substrate(s) | Change from baseline at two weeks on diet
  Change measured by respiratory exchange ratio (VCO2/VO2) difference between baseline and at two weeks on diet
Changes in blood glucose (mg/dL) | Change from baseline at two weeks on diet
  Change as measured by the difference between blood glucose levels at baseline and at week two on diet
Changes in ketone levels (mM or mcg/mL) | Change from baseline at two weeks on diet
  Change measured by the difference between ketone levels between baseline and at two weeks on diet
Changes in hemoglobin A1C (HbA1C) (%) | Change from baseline at two weeks on diet
  Change measured by the difference between A1C levels at baseline and at 2 weeks on diet
Changes in C-reactive protein (CRP) (mg/L) | Change from baseline at two weeks on diet
  Change measured by the difference between CRP levels at baseline and at 2 weeks on diet
Changes in lipid particle size (nm) | Change from baseline at two weeks on diet
  Change measured by the difference in lipid particle size at baseline and at 2 weeks on diet using Nuclear Magnetic Resonance (NMR).
Changes in lipid particle number (nmol/L and/or μmol/L) | Change from baseline at two weeks on diet
  Change measured by the difference in lipid particle number at baseline and at 2 weeks on diet using Nuclear Magnetic Resonance (NMR)
Changes in insulin sensitivity [(Homeostatic Model Assessment of Insulin Resistance (HOMA-IR score)] | Change from baseline at two weeks on diet
  Change as measured by the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) score using fasting insulin and glucose from longitudinal blood specimens at baseline and at two weeks on diet. The HOMA-IR test tests how resistant a participant is to insulin. A score of less than 1 indicates that a participant is insulin-sensitive, a score greater than 1.9 indicates some insulin resistance, and a score greater than 2.9 indicates significant insulin resistance.
Prostate health changes | Change from baseline at two weeks on diet
  As measured by changes in the Prostate Health Index
Safety and tolerability of the diets | Through study completion, an average of 7.5 month
  Safety and tolerability measured by the number of adverse events and by the gastric tolerance questionnaire
Changes in alpha and beta diversity of the gut microbiome | Change from baseline at two weeks on diet
  Changes measured by Shannon or Simpson diversity index (alpha diversity) and pairwise Bray-Curtis metric values (beta diversity)
Changes in dietary behavior | Through study completion, an average of 7.5 months
  Behavioral changes measured by validated 24 hour dietary recalls collected by trained dietetics personnel on 2 week days and 1 weekend to capture specific dietary information
Diet compliance | throughout controlled feeding period(s), two weeks per diet
  Compliance measured by >90% of provided calories consumed

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Weight, MD, Principal Investigator — Center Director, Cleveland Clinic Urologic Oncology
Locations (1):
- Case Comprehensive Cancer Center, Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Background] Freedland SJ, Howard L, Allen J, Smith J, Stout J, Aronson W, Inman BA, Armstrong AJ, George D, Westman E, Lin PH. A lifestyle intervention of weight loss via a low-carbohydrate diet plus walking to reduce metabolic disturbances caused by androgen deprivation therapy among prostate cancer patients: carbohydrate and prostate study 1 (CAPS1) randomized controlled trial. Prostate Cancer Prostatic Dis. 2019 Sep;22(3):428-437. doi: 10.1038/s41391-019-0126-5. Epub 2019 Jan 21. PMID 30664736
- [Background] Ornish D, Weidner G, Fair WR, Marlin R, Pettengill EB, Raisin CJ, Dunn-Emke S, Crutchfield L, Jacobs FN, Barnard RJ, Aronson WJ, McCormac P, McKnight DJ, Fein JD, Dnistrian AM, Weinstein J, Ngo TH, Mendell NR, Carroll PR. Intensive lifestyle changes may affect the progression of prostate cancer. J Urol. 2005 Sep;174(3):1065-9; discussion 1069-70. doi: 10.1097/01.ju.0000169487.49018.73. PMID 16094059